CLINICAL TRIAL: NCT00155662
Title: The Effect of a Work-hardening Program for Return-to-work for Workers With Low Back Pain
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: National Taiwan University Hospital (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None
Other Study IDs: 9100002906
Record Dates: First submitted 2005-09-09; First posted 2005-09-12 (Estimated); Last update posted 2012-12-06 (Estimated); Status verified 2012-12

CONDITIONS: Low Back Pain
Keywords: work hardening; chronic low back pain over 3 months
MeSH Terms: conditions — Low Back Pain

INTERVENTIONS:
Behavioral: work-hardening program

SUMMARY:
Occupational injury results in family economic crisis and national productivity loss; it is really becoming an important issue in Taiwanese society. Low back pain is the most frequent injury affecting workers. In addition to the prevention of injury, having a work-hardening program and getting the injured workers returned to work are also challenges for medical personnel. The purposes of this study are:

1. to develop a guideline to assess the low back pain workers' impairment and working capacity;
2. to formulate a feasible work-hardening program for the low back pain workers; and
3. to execute the program, evaluate the training effect and then follow up the rate of return to work of the low back pain workers.

In the first year, a guideline for assessment of low back impairment and working capacity will be developed. It may consist of the demographic data, the working status, the physical need in work, trunk muscle isokinetic strength, Oswestry low back disability questionnaire, functional capacity evaluation and quality of life questionnaire. The whole assessment package will be empirically applied in low back pain workers and the validity and reliability will be tested. A work-hardening program for low back pain workers will be established in the first year through meetings with experts and literature review. The work-hardening program will consist of training of trunk muscle strength, flexibility, and general fitness. A sling-exercise training model will be applied in the program. In the second year, low back pain workers in outpatient departments will be recruited with their own agreement and grouped randomly into either the work-hardening group or the control group. The expected number of subjects is 30 in each group. According to the result of impairment assessment and work capacity, the workers in the work-hardening group will start the individualized work-hardening program for 3 months. After the program, the workers will be assessed again to evaluate the training's effect, and the investigators will follow the rate of return to work among them 3 and 6 months after the program. The workers in the control group will be followed for 6 and 9 months after enrollment to collect the rate of return to work in this group.

DETAILED DESCRIPTION:
Occupational injury results in family economic crisis and national productivity loss; it is really becoming an important issue in our society. Low back pain is the most frequent injury affecting workers. In addition to the prevention of injury, having a work-hardening program and getting the injured workers returned to work are also challenges for medical personnel. The purposes of this study are:

1. to develop a guideline to assess the low back pain workers' impairment and working capacity;
2. to formulate a feasible work-hardening program for the low back pain workers; and
3. to execute the program, evaluate the training effect and then follow up the rate of return to work of the low back pain workers.

In the first year, a guideline for assessment of low back impairment and working capacity will be developed. It may consist of the demographic data, the working status, the physical need in work, trunk muscle isokinetic strength, Oswestry low back disability questionnaire, functional capacity evaluation and quality of life questionnaire. The whole assessment package will be empirically applied in low back pain workers and the validity and reliability will be tested. A work-hardening program for low back pain workers will be established in the first year through meetings and literature review. The work-hardening program will consist of training of trunk muscle strength, flexibility, and general fitness. A sling-exercise-training model will be applied in the program. In the second year, low back pain workers in outpatient departments will be recruited with their own agreement and grouped randomly into either the work-hardening group or the control group. The expected number of subjects is 30 in each group. According to the result of impairment assessment and work capacity, the workers in the work-hardening group will start the individualized work-hardening program for 3 months. After the program, the workers will be assessed again to evaluate the training's effect, and the investigators will follow the rate of return to work among them 3 and 6 months after the program. The workers in the control group will be followed for 6 and 9 months after enrollment to collect the rate of return to work in this group.

ELIGIBILITY:
Inclusion Criteria:

* Aged 18 to 65 years
* Have a job
* Low back pain

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2002-08; Primary Completion 2004-12 (Actual); Study Completion 2007-09 (Actual)

PRIMARY OUTCOMES:
functional capacity evaluation, Oswestry disability index

SECONDARY OUTCOMES:
low back pain, work hardening

CONTACTS AND LOCATIONS:
Overall Officials: J Y Tsauo, PhD, Study Director — Grad School of PT, College of Medicine, NTU
Locations (1):
- National Taiwan University Hospital, Taipei, Taiwan